CLINICAL TRIAL: NCT02396745
Title: A Prospective Feasibility Study to Evaluate the Safety and Efficacy of Transoral Endoscopic Circumferential Esophageal Resection With Extracellular Matrix (ECM) Placement to Treat Barrett's Esophagus With High-grade Dysplasia (HGD)
Brief Title: TECR & ECM Placement for Esophageal High Grade Dysplasia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Serious Adverse Event of Patient who completed study and follow-up.
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Collaborators: Integra LifeSciences Corporation (Industry)
Responsible Party: Principal Investigator, Blair Jobe, MD, Director, Esophageal and Lung Institute, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-024
Record Dates: First submitted 2015-03-19; First posted 2015-03-24 (Estimated); Results first posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-02

CONDITIONS: Barrett Esophagus; Esophagus; High Grade Dysplasia
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (1):
- TECR & ECM (Experimental): Subjects undergoing TECR with ECM placement Intervention is Trans-oral Endoscopic circumferential resection (TECR) with placement of extra-cellular matrix (ECM)
  Interventions: Device: Subjects undergoing TECR with ECM placement (ACell MatriStem, Boston Scientific WallFlex))

INTERVENTIONS:
Device: Subjects undergoing TECR with ECM placement (ACell MatriStem, Boston Scientific WallFlex)) — TECR will be performed to resect the entire length and area of BE lesion.
  ECM PLACEMENT:
  Following resection, the exposed area will be covered with a 6 ply sheet of ACell MatriStem® Surgical Matrix PSMX ECM (ACell Inc., Columbia, MA). The ECM will be placed and held in position for 14 days (±4 days) using a Boston Scientific WallFlex™ Fully Covered Esophageal Stent (Boston Scientific, Boston, MA).
  Other Names: ACell, Inc. MatriStem® Surgical Matrix PSMX; Boston Scientific, WallFlex™ Fully Covered Esophageal Stent

SUMMARY:
This study will test the safety and effectiveness of esophageal transoral endoscopic circumferential resection (TECR) using an extracellular matrix (ECM) placement to treat Barrett's esophagus in patients with high-grade dysplasia (HGD). Endoscopic circumferential resection using ECM placement has been introduced as a less invasive, externally incision-less approach to treat patients with esophageal high grade dysplasia; a pre-cancerous condition. In this procedure, the entire length of diseased (abnormal) mucosa (esophagus lining) will be removed using an endoscope that will be inserted through the mouth. The ECM will be placed over the area that is being removed with a temporary, expandable stent to prevent narrowing of the esophagus. The stent is being used to hold the ECM in place as the body begins the healing process. This stent will be removed 14 days (±4 days) after this procedure. Follow-up esophagogastroduodenoscopies (EGD), barium swallow x-ray tests, and questionnaires will take place for 12 months following the procedure. The result of this study may help doctors determine if this procedure would be a more effective treatment option for HGD in the future.

DETAILED DESCRIPTION:
This is a single-center, prospective, single arm study involving 10 patients with an established diagnosis of Barrett's Esophagus (BE) with High Grade Dysplasia (HGD). Potential subjects will be prescreened to assess eligibility and must meet inclusion criteria. In order to make this initial qualification, pathology results of biopsies and EMR collected during initial EGD will be made available to the Investigator prior to patient consent. Following informed consent and as part of routine care, all potential participants will undergo endoscopic ultrasound (EUS) and a PET/CT scan to confirm that there is no lymph node involvement or other metastatic lesions prior to the procedure. Clinical data will be collected at baseline to assess the subjects' medical status including: demographics, medical history, physical examination, vital signs, and blood testing. Cardiac and pulmonary clearance will be obtained if needed based on medical history and will include a chest x-ray, ECG, and pulmonary function test. In addition, the subjects will complete three questionnaires prior to the procedure: dysphagia severity questionnaire, SF-36, and GERD-HRQL.

At the time of the procedure, participants will undergo TECR with ECM placement using a fully covered self-expanding metal stent to temporarily hold the ECM in place. Prior to hospital discharge, a barium swallow test (BaSW) will be performed at Day 1 following the study procedure to evaluate the passage of contrast through the GEJ. If the BaSW results in suspicious findings of esophageal perforation or mucosal necrosis, an upper endoscopy will be performed for further evaluation. The first primary safety endpoint for this study will be assessed following the procedure and BaSW and before discharge from the hospital. At this time point any adverse events will be assessed and recorded.

All subjects will undergo the same follow-up procedures, including questionnaires and post-procedure EGDs performed at Week 2, Month 1, Month 3, Month 6, Month 9 and Month 12 to visually assess tissue healing, recurrent disease, and if stricture formation is present. Biopsies will be taken during follow-up EGDs so that pathology can rule out recurrence of BE and HGD. Subjects will have a barium swallow x-ray at Month 1, Month 3, Month 6, Month 9, and Month 12 to evaluate the potential presence of stricture formation.

During Week 2 EGD, the stent will be removed during the upper endoscopy. If at any time point a subject has dysphagia with stricture formation (30% reduction in esophageal luminal diameter), routine dilation using a balloon catheter will be performed during the EGD. Validated questionnaires including dysphagia severity questionnaire, SF-36 and GERD-HRQL will be administered to objectively assess the severity of symptoms and quality of life based upon self-reported data. Additionally, adverse events will be assessed and recorded at all follow-up time points.

After completion of the Month 12 visit, subjects will be followed on a routine care basis at the Esophageal & Lung Institute.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age and no more than 80 years of age.
2. Have an established diagnosis of HGD

   a. Specific diagnosis and grading will be determined by pathology review of biopsy tissue collected during baseline EGD as part of a patient's standard of care.
3. Have no evidence of lymphovascular invasion.
4. Have no lymph node or other metastatic involvement based on EUS and FDG-PET/CT.
5. Diameter of affected tissue must warrant circumferential excision a. Subjects must have biopsy confirmed HGD in three of four esophageal quadrants at two levels spaced two centimeters apart (minimum of 6/8 biopsies indicating HGD). If two biopsies are normal (contain no HGD) they must be located on separate levels in two different quadrants.

5. Must be an appropriate or reasonable surgical candidate. 6. Have demonstrated an understanding and signed an approved informed consent form for participation in this study.

Exclusion Criteria:

1. Have lesions into or deeper than mucosal layer (superficial (T1a) Esophageal adenocarcinoma).

   a. Those requiring endoscopic submucosal dissection (ESD) are not eligible for this study
2. Have presence of lymphovascular invasion.
3. Require resection length longer than 10 cm.
4. Have any lymph node or other metastatic involvement based on EUS and FDG-PET/CT.
5. Have history of any kind of previous esophageal surgery (i.e. anti-reflux surgery).
6. Are pregnant or planning to become pregnant.
7. Have coagulation disorders.
8. Have a known hypersensitivity to porcine-based materials.
9. Have an uncontrolled comorbid medical condition that would adversely affect participation in the trial.
10. Has a clinically significant psychological illness that in the physician's opinion would prohibit the subject's ability to meet the protocol requirements.
11. Are unable or unwilling to provide informed consent and/or fulfill the protocol follow-up requirements.

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-03-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- West Penn Allegheny Health System, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rice TW, Zuccaro G Jr, Adelstein DJ, Rybicki LA, Blackstone EH, Goldblum JR. Esophageal carcinoma: depth of tumor invasion is predictive of regional lymph node status. Ann Thorac Surg. 1998 Mar;65(3):787-92. doi: 10.1016/s0003-4975(97)01387-8. PMID 9527214
- [Background] Witteman BP, Foxwell TJ, Monsheimer S, Gelrud A, Eid GM, Nieponice A, O'Rourke RW, Hoppo T, Bouvy ND, Badylak SF, Jobe BA. Transoral endoscopic inner layer esophagectomy: management of high-grade dysplasia and superficial cancer with organ preservation. J Gastrointest Surg. 2009 Dec;13(12):2104-12. doi: 10.1007/s11605-009-1053-x. Epub 2009 Oct 14. PMID 19826883
- [Background] Badylak SF, Vorp DA, Spievack AR, Simmons-Byrd A, Hanke J, Freytes DO, Thapa A, Gilbert TW, Nieponice A. Esophageal reconstruction with ECM and muscle tissue in a dog model. J Surg Res. 2005 Sep;128(1):87-97. doi: 10.1016/j.jss.2005.03.002. PMID 15922361
- [Background] Nieponice A, Gilbert TW, Badylak SF. Reinforcement of esophageal anastomoses with an extracellular matrix scaffold in a canine model. Ann Thorac Surg. 2006 Dec;82(6):2050-8. doi: 10.1016/j.athoracsur.2006.06.036. PMID 17126109
- [Background] Nieponice A, McGrath K, Qureshi I, Beckman EJ, Luketich JD, Gilbert TW, Badylak SF. An extracellular matrix scaffold for esophageal stricture prevention after circumferential EMR. Gastrointest Endosc. 2009 Feb;69(2):289-96. doi: 10.1016/j.gie.2008.04.022. Epub 2008 Jul 26. PMID 18657808
- [Background] Badylak SF, Hoppo T, Nieponice A, Gilbert TW, Davison JM, Jobe BA. Esophageal preservation in five male patients after endoscopic inner-layer circumferential resection in the setting of superficial cancer: a regenerative medicine approach with a biologic scaffold. Tissue Eng Part A. 2011 Jun;17(11-12):1643-50. doi: 10.1089/ten.TEA.2010.0739. Epub 2011 Mar 28. PMID 21306292
- [Background] Hoppo T, Badylak SF, Jobe BA. A novel esophageal-preserving approach to treat high-grade dysplasia and superficial adenocarcinoma in the presence of chronic gastroesophageal reflux disease. World J Surg. 2012 Oct;36(10):2390-3. doi: 10.1007/s00268-012-1698-6. PMID 22736346
- [Background] Buscaglia JM, Ho S, Sethi A, Dimaio CJ, Nagula S, Stavropoulos SN, Gonda TA, Poneros JM, Stevens PD. Fully covered self-expandable metal stents for benign esophageal disease: a multicenter retrospective case series of 31 patients. Gastrointest Endosc. 2011 Jul;74(1):207-11. doi: 10.1016/j.gie.2011.02.024. Epub 2011 May 6. No abstract available. PMID 21549373
- [Background] Liu J, Hu Y, Cui C, Li Y, Lin X, Fu J. Removable, fully covered, self-expandable metal stents for the treatment of refractory benign esophagogastric anastomotic strictures. Dysphagia. 2012 Jun;27(2):260-4. doi: 10.1007/s00455-011-9361-1. Epub 2011 Aug 9. PMID 21826422
- [Background] Bakken JC, Wong Kee Song LM, de Groen PC, Baron TH. Use of a fully covered self-expandable metal stent for the treatment of benign esophageal diseases. Gastrointest Endosc. 2010 Oct;72(4):712-20. doi: 10.1016/j.gie.2010.06.028. PMID 20883848
- [Background] Eloubeidi MA, Lopes TL. Novel removable internally fully covered self-expanding metal esophageal stent: feasibility, technique of removal, and tissue response in humans. Am J Gastroenterol. 2009 Jun;104(6):1374-81. doi: 10.1038/ajg.2009.133. Epub 2009 Apr 28. PMID 19491851
- [Background] Yoon CJ, Shin JH, Song HY, Lim JO, Yoon HK, Sung KB. Removal of retrievable esophageal and gastrointestinal stents: experience in 113 patients. AJR Am J Roentgenol. 2004 Nov;183(5):1437-44. doi: 10.2214/ajr.183.5.1831437. PMID 15505317
- [Background] Baron TH, Burgart LJ, Pochron NL. An internally covered (lined) self-expanding metal esophageal stent: tissue response in a porcine model. Gastrointest Endosc. 2006 Aug;64(2):263-7. doi: 10.1016/j.gie.2006.03.936. PMID 16860080
- [Background] Sharma P, Kozarek R; Practice Parameters Committee of American College of Gastroenterology. Role of esophageal stents in benign and malignant diseases. Am J Gastroenterol. 2010 Feb;105(2):258-73; quiz 274. doi: 10.1038/ajg.2009.684. Epub 2009 Dec 22. PMID 20029413
- [Background] Hirdes MM, Siersema PD, Houben MH, Weusten BL, Vleggaar FP. Stent-in-stent technique for removal of embedded esophageal self-expanding metal stents. Am J Gastroenterol. 2011 Feb;106(2):286-93. doi: 10.1038/ajg.2010.394. Epub 2010 Oct 12. PMID 20940709
- [Background] van Heijl M, Gooszen JA, Fockens P, Busch OR, van Lanschot JJ, van Berge Henegouwen MI. Risk factors for development of benign cervical strictures after esophagectomy. Ann Surg. 2010 Jun;251(6):1064-9. doi: 10.1097/SLA.0b013e3181deb4b7. PMID 20485137

RESULTS

PARTICIPANT FLOW:
Groups:
- TECR & ECM: Subjects undergoing TECR with ECM placement Intervention is Trans-oral Endoscopic circumferential resection (TECR) with placement of extra-cellular matrix (ECM)
  Subjects undergoing TECR with ECM placement (ACell MatriStem, Boston Scientific WallFlex)): TECR will be performed to resect the entire length and area of BE lesion.
  ECM PLACEMENT:
  Following resection, the exposed area will be covered with a 6 ply sheet of ACell MatriStem® Surgical Matrix PSMX ECM (ACell Inc., Columbia, MA). The ECM will be placed and held in position for 14 days (±4 days) using a Boston Scientific WallFlex™ Fully Covered Esophageal Stent (Boston Scientific, Boston, MA).
Period: Overall Study
Arm/Group | TECR & ECM
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TECR & ECM
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants] — Between 18 and 80 years
  Participants
    <=18 years | 0
    Between 18 and 65 years | 0
    >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Stricture Formation
Description: To evaluate incidence of stricture formation requiring dilation (≥30% luminal diameter reduction with dysphagia) following TECR with ECM placement. Evidence of stricture formation will be confirmed endoscopically at 2 weeks, and endoscopically and through barium swallow at Month 1, Month 3, Month 6, Month 9, and Month 12 post procedure, and the proportion of subjects with and without stricture formation at the trial endpoints will be compared to historical data.
Time Frame: 12 months following procedure
Population: Study terminated early. Subject participant experienced SAE and was followed for safety, no data outcomes analyzed
Arm/Group | TECR & ECM
Number analyzed (Participants) | 0

2. Primary Outcome: Efficacy: Recurrent Disease
Description: To evaluate incidence of recurrence of BE with HGD through 12 months following TECR with ECM placement. Incidence of disease recurrence will be confirmed endoscopically with pathology confirmed biopsies at 2 weeks, Month 1, Month 3, Month 6, Month 9, and Month 12 post procedure, and the proportion of subjects with and without disease recurrence at the trial endpoints will be compared to historical data.
Time Frame: 12 months following procedure
Population: Study terminated early. Subject participant experienced SAE and was followed for safety, no data outcomes analyzed
Arm/Group | TECR & ECM
Number analyzed (Participants) | 0

3. Primary Outcome: Safety: Acute (Serious System and Procedure Related Adverse Events)
Description: To demonstrate the acute safety of TECR with ECM placement for treatment of BE with HGD by evaluating all serious system and procedure related adverse events occurring in the first 2 weeks post procedure.
Time Frame: Two weeks following procedure
Measure: Count of Participants; unit: Participants
Arm/Group | TECR & ECM
Number analyzed (Participants) | 1
Participants | 1

4. Primary Outcome: Safety: Long-term (Study Related Adverse Events)
Description: To demonstrate the long-term safety of TECR with ECM placement for treatment of BE with HGD by evaluating all study related adverse events occurring more than 2 weeks post procedure through 12 months post procedure.
Time Frame: Two weeks through 12 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | TECR & ECM
Number analyzed (Participants) | 1
Participants | 1

5. Secondary Outcome: Stent Migration
Description: To record the incidence of stent migration at 2 weeks post procedure. Stent migration will be determined endoscopically, and defined as any movement from initial deployment location greater than 1cm.
Time Frame: 2 weeks
Population: Study terminated early. Subject participant experienced SAE and was followed for safety, no data outcomes analyzed
Arm/Group | TECR & ECM
Number analyzed (Participants) | 0

6. Secondary Outcome: Stent Integrity (e.g. Stent Fracture)
Description: To record incidences of poor stent integrity during removal (e.g. stent fracture).
Time Frame: 2 weeks
Population: Study terminated early. Subject participant experienced SAE and was followed for safety, no data outcomes analyzed
Arm/Group | TECR & ECM
Number analyzed (Participants) | 0

7. Secondary Outcome: Additional Interventions (Number of Subsequent Follow up Treatment Interventions)
Description: To record the number of subsequent follow up treatment interventions (aside from study-related follow up time points) required post-procedure through 12 months.
Time Frame: 12 months
Population: Study terminated early. Subject participant experienced SAE and was followed for safety, no data outcomes analyzed
Arm/Group | TECR & ECM
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year, 10 months
Arm/Group | TECR & ECM
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TECR & ECM (N=1)
Dysphagia (Gastrointestinal disorders) | 1 (20) — Dysphagia due to stricture from stent migration
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TECR & ECM (N=1)
Dysphagia (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT02396745/Prot_SAP_000.pdf